CLINICAL TRIAL: NCT02924987
Title: Effect of Aflibercept (Eylea®) in the Management of Bevacizumab (Avastin®) Resistant Diabetic Macular Edema
Acronym: Eylea
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Flavio Rezende, Principal Investigator, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hôpital Maisonneuve-Rosemont
Record Dates: First submitted 2016-01-12; First posted 2016-10-05 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aflibercept injection (Other): Not applicable. There will be no randomization nor stratification to any to study arms or groups.
  Interventions: Drug: Aflibercept Injection

INTERVENTIONS:
Drug: Aflibercept Injection — Intravitreal injections of 0.05 mL (2mg) of Aflibercept will be injected. The intravitreal between the first 5 treatments sessions is 4 weeks, and the interval for the following treatment sessions up to week 52 is 8 weeks.
  Other Names: Eylea

SUMMARY:
Multicenter randomized trials have demonstrated the safety and efficacy of intravitreal anti-vascular endothelial growth factor (anti-VEGF) agents for the treatment of diabetic macular edema. The results are generally good in the short term, with approximately 75% of patients maintaining or improving vision after initiation of treatment. Despite this favorable outcome, the observation of persistent fluid is not infrequent during treatment, even in patients undergoing monthly treatment sessions. Persistent fluid was observed on optical coherence tomography (OCT) in 70.9% of patients receiving bevacizumab monthly and in 79% of those receiving bevacizumab as needed at the end of the first year in the Comparison of diabetic macular edema. Treatment Trials. It is possible that resolution of this fluid, especially when it is centrally located (i.e., foveal), might result in better visual outcomes.

A drug with higher VEGF-binding affinity may help patients with persistent fluid despite treatment with bevacizumab. Aflibercept is a new intravitreal VEGF antagonist approved on 28 November 2014 by the Health Canada for the treatment of diabetic macular edema.

In contrast to the antibody-based VEGF binding strategy used by bevacizumab, aflibercept incorporates the second binding domain of the VEGFR-1 receptor and the third domain of the VEGFR-2 receptor. By fusing these extracellular protein sequences to the Fc segment of a human IgG backbone, developers have created a chimeric protein with a very high VEGF binding affinity. Aflibercept binds all isomers of the VEGF-A family like bevacizumab, but it also binds VEGF-B and placental growth factors 1 and 2,1,2 which have been both implicated in the pathogenesis of diabetic retinopathy and of age-related macular degeneration. In addition, because of the increased trough binding activity and the stronger binding affinity, aflibercept should be efficacious in neutralizing VEGF more effectively and for longer duration.

DETAILED DESCRIPTION:
In this study patients recruitment, clinical care and follow-up will be conducted by:

Dr Flavio Rezende: Principal-Investigator and Dr Radwan Ajlan: Co-Investigator.

1. Purpose: To evaluate the visual acuity outcomes and macular changes at 6 and 12 months of intravitreal aflibercept (2.0 mg) in eyes with persistent center involved diabetic macular edema despite intravitreal bevacizumab therapy.
2. Overall Goal of Study: The goal of this study is to evaluate the effect of aflibercept on macular edema in patients with diabetic macular edema resistant to bevacizumab.
3. Specific objectives: To evaluate the visual acuity outcomes and macular changes after 6 and 12 months of intravitreal aflibercept (2.0 mg) in eyes with persistent foveal fluid secondary to diabetic macular edema despite previous optimum gold standard therapy with intravitreal bevacizumab. More specifically, to assess:

   * Mean change in central subfield thickness (CST) from baseline, 6 month after switching to aflibercept.
   * Mean change in CST from baseline, 12 months after switching to aflibercept.
   * Mean change in best corrected visual acuity (BCVA) from baseline, 6 months after switching to aflibercept.
   * Mean change in BCVA from baseline, 12 months after switching to aflibercept
4. Study Design: Phase 4 open label clinical trial. Intravitreal injection of 0.05 mL (2mg) of aflibercept will be injected. The intravitreal between the first 5 treatments sessions is 4 weeks, and the intravitreal for the following treatment sessions up to week 52 is 8 weeks.
5. Subjects: 40 patients seen in the retinal clinic of the Hospital Maisonneuve-Rosemont with foveal fluid secondary to diabetic macular edema despite previous optimum gold standard therapy with intravitreal bevacizumab will be assessed for eligibility.

ELIGIBILITY:
Inclusion Criteria:

* Eyes to be included in the series must have had at least six consecutive monthly intravitreal injections of bevacizumab for the treatment of diabetic macular edema and presented tomographic signals suggestive of foveal fluid on spectral-domain optical coherence tomography (SD-OCT) 4 weeks after the last treatment session. The interval between each of the last 3 consecutive bevacizumab treatments and the interval between the last bevacizumab and the SD-OCT imaging not exceeding 37 days.
* Persistent foveal fluid is defined as the observation of hypo-reflective spaces on OCT at the fovea (fovea centralis), which measures approximately 1.5 mm (1500 μm) or one disc diameter in size centered at the macular umbo. Tomographic changes will be measured by SD-OCT using the macular thickness maps.
* BCVA must be better than 20/800. Only 1 eye from each patient will be included in the study. If both eyes are affected, the better seeing eye will be included, since no previous meaningful difference was found in patients with 20/40 or better when treated with bevacizumab or aflibercept.3

Exclusion Criteria:

* An ocular media opacity that might interfere with visual acuity, assessment of toxicity, or photographic fundus documentation of the macular area.
* A history of vitrectomy.
* Known coagulation abnormalities, stroke, or recurrent use of anticoagulative medication other than aspirin.
* Pregnancy, or planning for pregnancy during the study time frame or the following 3 months.
* Patients actively undergoing other ocular treatment options such as topical nonsteroidal anti-inflammatory drugs NSAIDs, topical steroids, or intravitreal steroids injections will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Macular central subfield thickness in micrometers | 6 Months
  Central subfield thickness in micrometers at 6 months measured by optical coherence tomography in micrometers (HRT+OCT Spectralis model, Heidelberg Engineering, Heidelberg, Germany).

SECONDARY OUTCOMES:
Macular central subfield thickness in micrometers at 12 months measured by optical coherence tomography in micrometers (HRT+OCT Spectralis model, Heidelberg Engineering, Heidelberg, Germany) | 12 months
Best corrected visual acuity at 12 months measured in letters using ETDRS chart | 12 months
Best corrected visual acuity at 6 months measured in letters using ETDRS chart | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Rezende, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- Maisonneuve Rosemont Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No